CLINICAL TRIAL: NCT04435795
Title: Ciclesonide Clinical Trial for COVID-19 Treatment
Brief Title: Inhaled Ciclesonide for Outpatients With COVID19
Acronym: CONTAIN
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: could not meet target enrolment
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Nicole Ezer, MD, FRCPC, MPH, Assistant Professor of Medicine, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-6696
Record Dates: First submitted 2020-06-16; First posted 2020-06-17 (Actual); Results first posted 2022-04-29 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-05

CONDITIONS: COVID 19
MeSH Terms: conditions — COVID-19 | interventions — ciclesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ciclesonide inhaled and nasal (Active Comparator): Intranasal ciclesonide BID 50mcg BID to each nostril and inhaled ciclesonide 600mcg BID x 14 days
  Interventions: Drug: Ciclesonide; Drug: Ciclesonide nasal
- Placebo (Placebo Comparator): Normal Saline intranasal BID and Placebo 3 puff MDI inhaled BID
  Interventions: Drug: Normal Saline intranasal and placebo inhaler

INTERVENTIONS:
Drug: Normal Saline intranasal and placebo inhaler — Normal Saline intranasal BID and Placebo 3 puff MDI inhaled BID
  Arms: Placebo
Drug: Ciclesonide — Ciclesonide 600mcg BID inhaled with aero chamber
  Other Names: Alvesco
  Arms: Ciclesonide inhaled and nasal
Drug: Ciclesonide nasal — intranasal ciclesonide 200 mcg DIE
  Other Names: Omnaris
  Arms: Ciclesonide inhaled and nasal

SUMMARY:
The CONTAIN (CiclesOnide cliNical TriAl covId-19 treatmeNt) is a randomized control study of ciclesonide vs placebo for mild covid-19 disease. The need for potential therapy for COVID-19 patients is urgent. Ciclesonide has shown encouraging in vitro results, is easy to be used and is readily available. It has a low rate of side effects and few interactions with other drugs. It is unusual to use an inhaled steroid drug for COVID-19 but there has been new data suggesting steroids may have an antiviral effect in addition to an anti-inflammatory effect. Investigators propose to use inhaled and nasal ciclesonide to stop viral replication in the nose and airways. Investigators hope this will accelerate recovery from COVID-19 illness in individuals who are not admitted to hospital at time of diagnosis of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

Symptomatic adult patients positive by PCR for COVID-19 within 5 days of enrollment with fever, cough, or shortness of breath. Provision of Informed Consent

At day 0, patients should be at home

Exclusion Criteria:

* Already on inhaled corticosteroid medication
* Currently using systemic steroids (oral or intravenous or intramuscular such as Prednisone) or use of steroids 7 days prior to enrolment
* Severely ill patients at enrollment (i.e., admitted to ICU at admission)
* Unable to self-administer the inhaler
* Known or suspected pregnancy and breastfeeding
* Known allergy to study medication or its components (non-medicinal ingredients; including lactose allergy (type I))
* Patients with untreated fungal, bacterial, or tubercular infections of the respiratory tract
* Current hospitalization
* Current use of oxygen at home or in the hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-07-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - University of British Columbia, Vancouver, British Columbia
  - Sunnybrook Hospital, Toronto, Ontario
  - McGill University Health Center, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ezer N, Belga S, Daneman N, Chan A, Smith BM, Daniels SA, Moran K, Besson C, Smyth LY, Bartlett SJ, Benedetti A, Martin JG, Lee TC, McDonald EG. Inhaled and intranasal ciclesonide for the treatment of covid-19 in adult outpatients: CONTAIN phase II randomised controlled trial. BMJ. 2021 Nov 2;375:e068060. doi: 10.1136/bmj-2021-068060. PMID 34728476
- See also: Trial website — https://contain-covid19.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolment to the trial began on 15 September 2020 in Quebec, 9 February 2021 in Ontario, and 22 March 2021 in British Columbia. The last participants were recruited on 8 June 2021.
Pre-assignment Details: Overall, 215 participants were randomised, and the modified intention-to-treat population included 203 adults with respiratory symptoms or fever.
Period: Overall Study
Arm/Group | Ciclesonide Inhaled and Nasal | Placebo
Started | 108 | 107
Completed | 105 | 98
Not Completed | 3 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ciclesonide Inhaled and Nasal | Placebo | Total
Number analyzed (Participants) | 105 | 98 | 203
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 35 [27 to 47] | 35 [27 to 45] | 35 [27 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 55 | 109
  Male | 51 | 43 | 94
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: African canadian | 3 | 2 | 5
  Ethnicity: Asian | 18 | 16 | 34
  Ethnicity: White | 63 | 53 | 116
  Ethnicity: Hispanic or Latino | 6 | 7 | 13
  Ethnicity: Middle Eastern | 6 | 12 | 18
  Ethnicity: South Asian | 6 | 6 | 12
  Ethnicity: Other | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  Canada: British Columbia | 51 | 51 | 102
  Canada: Ontario | 19 | 13 | 32
  Canada: Quebec | 35 | 34 | 69

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With no Symptoms of Cough, Fever or Dyspnea
Description: Proportion of participants with no symptoms of cough, fever or dyspnea at day 7
Time Frame: day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Ciclesonide Inhaled and Nasal | Placebo
Number analyzed (Participants) | 105 | 98
Participants | 42 | 34

2. Secondary Outcome: Proportion of Participants With no Symptoms of Cough, Fever or Dyspnea
Description: Proportion of participants with no symptoms of cough, fever or dyspnea at Day 14
Time Frame: Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Ciclesonide Inhaled and Nasal | Placebo
Number analyzed (Participants) | 105 | 98
Participants | 95 | 91

3. Secondary Outcome: Overall Feeling: Proportion Who Are Reporting That They Are "Very Much Improved" or "Much Improved" at Day 7
Description: Proportion who are reporting that they are "very much improved" or "much improved"
Time Frame: Day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Ciclesonide Inhaled and Nasal | Placebo
Number analyzed (Participants) | 105 | 98
Participants | 77 | 74

4. Secondary Outcome: Overall Feeling: Proportion Who Are Reporting That They Are "Very Much Improved" or "Much Improved" at Day 14
Description: Proportion who are reporting that they are "very much improved" or "much improved"
Time Frame: Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Ciclesonide Inhaled and Nasal | Placebo
Number analyzed (Participants) | 105 | 98
Participants | 95 | 91

5. Secondary Outcome: Improvement in Dyspnea: Resolution of Dyspnea at Day 7
Description: Dyspnea was defined as reporting "shortness of breath" or "chest congestion" or "chest tightness". In those who reported dyspnea at baseline, resolution will be defined as having no symptoms in these three areas.
Time Frame: day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Ciclesonide Inhaled and Nasal | Placebo
Number analyzed (Participants) | 53 | 49
Participants | 38 | 27

6. Secondary Outcome: Improvement in Cough at Day 7: Proportion of Patient With a Reduction of Cough Symptoms at Day 7
Description: Improvement of wet or dry cough. Analysis limited to patients who reported cough at baseline. Defined as a 2 point decrease, or a decrease to 0 on a visual analogue scale that ranged from 0 for no symptoms to 10 for severe symptoms
Time Frame: day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Ciclesonide Inhaled and Nasal | Placebo
Number analyzed (Participants) | 89 | 86
Participants | 57 | 54

7. Secondary Outcome: Proportion of Participants Hospitalized for SARS-CoV-2
Description: Hospitalization for SARS-CoV-2 related illness
Time Frame: day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Ciclesonide Inhaled and Nasal | Placebo
Number analyzed (Participants) | 105 | 98
Participants | 6 | 3

8. Secondary Outcome: Mortality
Description: All cause mortality
Time Frame: day 29
Measure: Count of Participants; unit: Participants
Arm/Group | Ciclesonide Inhaled and Nasal | Placebo
Number analyzed (Participants) | 105 | 98
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 29 Days
Arm/Group | Ciclesonide Inhaled and Nasal | Placebo
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/98
Serious Adverse Events (participants affected / at risk) | 7/105 | 5/98
Other Adverse Events (participants affected / at risk) | 23/105 | 15/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ciclesonide Inhaled and Nasal (N=105) | Placebo (N=98)
Hospithalization (Respiratory, thoracic and mediastinal disorders) | 6 | 3 — SAE related to COVID-19, not to the study drug
Visit to the emergency department (Respiratory, thoracic and mediastinal disorders) | 1 | 3 — Related to COVID-19, not to the study drug
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ciclesonide Inhaled and Nasal (N=105) | Placebo (N=98)
Thrush (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Severe headache (General disorders) | 13 | 5
Voice change (General disorders) | 2 | 2
throat irritaiton (General disorders) | 7 | 5
Dry mouth (General disorders) | 2 | 3
Dry nose, irritated nose or nosebleed (General disorders) | 4 | 1
Dizziness (General disorders) | 1 | 0
Nausea (General disorders) | 11 | 2
Wheeze (General disorders) | 0 | 1
Other (General disorders) | 6 | 3

LIMITATIONS AND CAVEATS:
We were unable to recruit the intended sample size given a rapid decline in cases of covid-19 in Canada following increases in vaccination.

In addition, we did not enrich the study population for older high risk people and cannot exclude a possible benefit in earlier symptom resolution and prevention of clinical deterioration in this group.

As our trial was stopped prematurely, we might have been underpowered to show a small benefit of ciclesonide on early symptom resolution

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/95/NCT04435795/Prot_SAP_000.pdf